CLINICAL TRIAL: NCT02974985
Title: A Study of the Lifting Capacity of Fillers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abington Memorial Hospital (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Allan Wulc, Allan E. Wulc, M.D., F.A.C.S, Abington Memorial Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-023
Record Dates: First submitted 2016-11-10; First posted 2016-11-29 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Esthetic & Topographic Shifts From Facial Fillers
Keywords: Facelift; HA Filler; Hyaluronic acid; Facial Rejuvenation; Aging Face; WIZDOM; Midface lift; Midface augmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- Women aged 40-50 (Experimental): Intervention--Injections of volumizing products Restylane L and Restylane Lyft with endpoint " a dramatic result is seen that is agreed upon by both subject and injector". The number of injections will be determined (and quantified) by both the patient and the PI to achieve this endpoint.
  Interventions: Device: injection of Restylane Lyft and Restylane L
- Women aged 50-60 (Experimental): Intervention--Injections of volumizing products Restylane L and Restylane Lyft with endpoint " a dramatic result is seen that is agreed upon by both subject and injector". The number of injections will be determined (and quantified) by both the patient and the PI to achieve this endpoint.
  Interventions: Device: injection of Restylane Lyft and Restylane L

INTERVENTIONS:
Device: injection of Restylane Lyft and Restylane L — Intervention--Injections of volumizing products to the midface, nasolabial fold, and marionette folds in female patients in two different age groups

SUMMARY:
Hyaluronic acid (HA) fillers are tested in-vitro to measure their lifting capacity, viscosity, cohesivity, and rheologic properties, and their lifting capacity has been tested in animal models. To date, there are no studies that measure the lifting capacity of fillers in an in-vivo human model.

The intention is to study the lifting capacity of fillers in a group of patients by comparing pre and post-procedure two and three-dimensional photographs using analytic software. Specifically, the PI is interested in determining the amount of tissue elevation created by injecting HAs Restylane-Lyft®, and Restylane-L® (Galderma Laboratories, L.P., Fort Worth, TX) to the midface and to the lower face, both in the anterior-posterior direction and in the vertical direction by using analytic software.

The research group has identified a reliable and reproducible quantitative assessment of midfacial position called WIZDOM (Width of the InterZygomatic Distance Of the Midface) to quantitatively evaluate the midface. It can be used as an objective tool to assess midfacial rejuvenation, whether with fat, fillers, or midface or facelift surgery. The Distance from WIZDOM to inner canthus, the WIZDOM -IC measurement increases with aging as the face deflates and descends, and, in the practice, is also a means of assessing the midface in youth and in aging. The PI's findings have been published in the Aesthetic Surgery Journal. The practice will also attempt to utilize this metric as a measure of midface aesthetic lifting capacity.

The practice will also employ 3 D photography and analytic software to determine degree of lift in mm in the y and z axis. (vertical and AP increase in dimension) pre and post- injection. (Vectra, Canfield, Fairfield, NJ)

We will recruit patients from a population of subjects that generally would receive fillers to improve changes associated with facial volume loss and divide them in to two groups based on chronologic age.

DETAILED DESCRIPTION:
All fillers will be injected in locations where the FDA has approved it for on-label indications (the cheek, subcutaneously and supraperiosteally, the dermis and subdermis for the correction of wrinkles and folds such as the nasolabial fold) and placed as usual and customary using techniques as practiced by the authors and as are accepted widely.

Additional steps prior to injection for this study are temporary sterile magic marker markings markers on the face and detailed photography, both 2D and 3D, that will be taken before, during, and after injection, and the segmentation of injections such that the midface will be injected prior to and separately from the lower face.

Three dimensional data will be analyzed using Vectra analytic software, and 2-D photographs will be analyzed by measuring improvements in WIZDOM (width of the interzygomatic distance of the midface) and its distance to the inner canthus.

ELIGIBILITY:
Inclusion Criteria:

* Women ages 40-60
* Midface, lower face volume loss and gravitational changes amenable to the administration of HA fillers.
* Filler requirements, based on experienced injector assessment, on the order of 8 syringes.

Exclusion Criteria:

* History of prior filler injections in the past 12 months.
* Pregnancy/planned pregnancy
* Allergy to HA products

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-09 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Degree and axes of volume shifts before and after injection of HA fillers | immediately after injection
  The investigators are using Vectra analysis software to analyze volume changes in 3D. dimensions after injection of hyaluronic acid filler.

SECONDARY OUTCOMES:
Measurement of MMVS | Two weeks post injections.
  Medicis Midface Volume Scale
Patient and Observer Satisfaction with Degree of Lift | immediately after injection
  Change in global aesthetic assessment measured from baseline.
Measure the capacity of fillers in the midface to change midface position. | immediately after injection
  H1 and Vectra analytic software: movement of measured points of reference on the face.
Measure the capacity of fillers in the midface to improve relationship between eyelid and cheek. | immediately after injection
  WIZDOM measurement and WIZDOM -IC measurement
Measure the capacity of fillers in the midface to change lower face position. | immediately after injection
  H1 and Vectra analytic software: movement of measured points of reference on the face.
Patient-reported subjective assessment of filler effect and satisfaction | Two weeks post injections.
  GAIS Scale
Investigator assessment of filler effect. | Two weeks post injections.
  GAIS scale

CONTACTS AND LOCATIONS:
Overall Officials: Allan E Wulc, M.D., Principal Investigator — Abington Hospital
Locations (1):
- W Cosmetic Surgery, Plymouth Meeting, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
will make protocols and statistics and photos available to all interested including esearch collaborators.

REFERENCES:
- [Background] Little JW. Volumetric perceptions in midfacial aging with altered priorities for rejuvenation. Plast Reconstr Surg. 2000 Jan;105(1):252-66; discussion 286-9. doi: 10.1097/00006534-200001000-00043. PMID 10626998
- [Background] Kablik J, Monheit GD, Yu L, Chang G, Gershkovich J. Comparative physical properties of hyaluronic acid dermal fillers. Dermatol Surg. 2009 Feb;35 Suppl 1:302-12. doi: 10.1111/j.1524-4725.2008.01046.x. PMID 19207319
- [Background] Swift A, Remington K. BeautiPHIcation: a global approach to facial beauty. Clin Plast Surg. 2011 Jul;38(3):347-77, v. doi: 10.1016/j.cps.2011.03.012. PMID 21824535
- [Background] Ramirez OM. Three-dimensional endoscopic midface enhancement: a personal quest for the ideal cheek rejuvenation. Plast Reconstr Surg. 2002 Jan;109(1):329-40; discussion 341-9. doi: 10.1097/00006534-200201000-00052. PMID 11786834
- [Background] Surek CC, Beut J, Stephens R, Jelks G, Lamb J. Pertinent anatomy and analysis for midface volumizing procedures. Plast Reconstr Surg. 2015 May;135(5):818e-829e. doi: 10.1097/PRS.0000000000001226. PMID 25919264
- [Background] Borrell M, Leslie DB, Tezel A. Lift capabilities of hyaluronic acid fillers. J Cosmet Laser Ther. 2011 Feb;13(1):21-7. doi: 10.3109/14764172.2011.552609. Epub 2011 Jan 21. PMID 21254807
- [Background] Pierre S, Liew S, Bernardin A. Basics of dermal filler rheology. Dermatol Surg. 2015 Apr;41 Suppl 1:S120-6. doi: 10.1097/DSS.0000000000000334. PMID 25828036
- [Background] Gold M. The science and art of hyaluronic acid dermal filler use in esthetic applications. J Cosmet Dermatol. 2009 Dec;8(4):301-7. doi: 10.1111/j.1473-2165.2009.00464.x. PMID 19958435
- [Background] Beer K, Lupo MP. Making the right choices: attaining predictable aesthetic results with dermal fillers. J Drugs Dermatol. 2010 May;9(5):458-65. PMID 20480788
- [Background] Carruthers J, Flynn TC, Geister TL, Gortelmeyer R, Hardas B, Himmrich S, Jones D, Kerscher M, de Maio M, Mohrmann C, Narins RS, Pooth R, Rzany B, Sattler G, Buchner L, Benter U, Breitscheidel L, Carruthers A. Validated assessment scales for the mid face. Dermatol Surg. 2012 Feb;38(2 Spec No.):320-32. doi: 10.1111/j.1524-4725.2011.02251.x. PMID 22316188
- [Background] Linkov G, Mally P, Czyz CN, Wulc AE. Quantification of the Aesthetically Desirable Female Midface Position. Aesthet Surg J. 2018 Feb 15;38(3):231-240. doi: 10.1093/asj/sjx122. PMID 29040391
- See also: Device Company website with FDA prescribing information and warnings — http://www.galderma.com